CLINICAL TRIAL: NCT03256474
Title: Can Community-acquired Bacterial Pneumonia in Children be Safely Managed Without Antibiotics in an Integrative Medicine Context? A Retrospective Cohort Analysis
Brief Title: Managing Bacterial Pneumonia in Children Without Antimicrobials
Status: Completed | Type: Observational
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: PKA_01
Record Dates: First submitted 2017-07-06; First posted 2017-08-22 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Combined Modality Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multimodal Therapy — Drugs, external applications like chest wraps, inhalations

SUMMARY:
Retrospective cohort analysis of children hospitalized for pneumonia comparing disease severity on admission, clinical course, treatment and outcomes and prospective telephone based Follow-Up assessement.

DETAILED DESCRIPTION:
The investigators will conduct a retrospective cohort analysis of children hospitalized for pneumonia at the Filderklinik between December 2006 and November 2010. The Bacterial Pneumonia Score, a validated composite laboratory, clinical and radiologic score developed by Moreno et al, will be retrospectively applied to define cases as either viral or bacterial pneumonia. The investigators will compare disease severity on admission, clinical course, and outcomes (in terms of complications, length of stay and readmission rates) between antimicrobial and non-antimicrobial managed bacterial pneumonia cases. Long-term Follow-Up will be assessed by telephone interviews with the parents.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission at the pediatric department of the Filderklinik.
* Admission diagnosis pneumonia (ICD J12.0, J12.1, J12.8, J12.9, J14, J15.1, J15.6, J15.7, J15.8, J15.9, J16.8, J18.0, J18.1, J18.8, J18.9 - all 12s, 15s, 16s, 18s)

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children from infancy till adolecence admitted to hospital (Filderklinik, Germany) for pneumonia treatment
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-02-25 (Actual)

PRIMARY OUTCOMES:
Cure rate of non-antimicrobial management of bacterial pneumonia | Between admission and 3 months after discharge
  Cure rate of non-antimicrobial management of bacterial pneumonia (in the following and in the final publication, the term "bacterial pneumonia" will be used for children who fulfill the Moreno criteria for pneumonia): % of children managed without antimicrobials since admission, without subsequent need for antimicrobials or readmission.
Medical complication rate | Between admission and 3 months after discharge
  Medical complication rate among children with bacterial pneumonia, treated with or without antimicrobials
Length of hospital stay | Between admission and 3 months after discharge
  Length of hospital stay for children with bacterial pneumonia, managed with or without antimicrobials
Readmission rate | 7 - 10 years after hospitalization
  Readmission rate for pneumonia among children with bacterial pneumonia, managed with or without antimicrobials
Temperature normalization | Between admission and 3 months after discharge
  Days to temperature normalization (< 38°C) in children with bacterial pneumonia, managed with or without antimicrobials
Days of supplemental oxygen need | Between admission and 3 months after discharge
  Days of supplemental oxygen need in children with bacterial pneumonia, managed with or without antimicrobials

SECONDARY OUTCOMES:
Changes in respiratory rate | Between admission and 3 months after discharge
  Changes in respiratory rate as an indicator for pulmonary infection
Changes in Bacterial Pneumonia Score | Between admission and 3 months after discharge
  Changes in Bacterial Pneumonia Score as an indicator for pulmonary infection
Changes in oxygen saturation | Between admission and 3 months after discharge
  Changes in oxygen saturation as an indicator for pulmonary infection
Changes in CRP | Between admission and 3 months after discharge
  Changes in CRP as an indicator for infection
Changes in leukocyte count | Between admission and 3 months after discharge
  Changes in leukocyte count as an indicator for infection
Changes in pH | Between admission and 3 months after discharge
  Changes in pH as an indicator for respiratory distress
Changes in pCO2 | Between admission and 3 months after discharge
  Changes in pCO2 as an indicator for respiratory distress
Rate of chronic and acute-infectious co-morbidities | Day of admission
  Rate of chronic and acute-infectious co-morbidities on admission in children with bacterial pneumonia, subsequently managed with or without antimicrobials
Utilization rate of a package of complementary treatment measures | Between admission and 3 months after discharge
  Utilization rate of a package of complementary treatment measures from anthroposophic medicine (including oral medications, inhalation and external nursing applications) in children managed with or without antimicrobials
Antimicrobial treatment rate in children with viral pneumonia | Between admission and 3 months after discharge
  Antimicrobial treatment rate in children classified as viral pneumonia by Bacterial Pneumonia Score
Number of patients treated with antipyretics | Between admission and 3 months after discharge
  Number of patients treated with antipyretics

CONTACTS AND LOCATIONS:
Locations (1):
- Arcim Institute, Filderstadt, Baden-Wurttemberg, Germany